CLINICAL TRIAL: NCT01064050
Title: Role of a Silicone Prosthesis to Prevent Airway Obstruction Recurrence After Therapeutic Bronchoscopy in Lung Cancers (SPOC Study)
Brief Title: Role of a Silicone Prosthesis to Prevent Airway Obstruction Recurrence in Lung Cancers
Acronym: SPOC
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulty to include patient
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Ministry of Health, France (Other Government); Ligue contre le cancer, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0708042; 2007-A01190-53 (Other: AFSSAPS)
Record Dates: First submitted 2010-02-02; First posted 2010-02-08 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Lung Neoplasm; Carcinoma, Non-Small-Cell Lung
Keywords: tumoral obstruction of the main stem bronchus; bronchoscopy; silicone stent
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- trachea-bronchial stent (Novatech) (Experimental)
  Interventions: Device: silicone trachea-bronchial stent Dumon (Novatech)
- control (No Intervention)

INTERVENTIONS:
Device: silicone trachea-bronchial stent Dumon (Novatech) — Bronchial desobstruction under interventional bronchoscopy, for inclusion, with the insertion of silicone stent trachea-bronchial covering the entire tumor area
  Arms: trachea-bronchial stent (Novatech)

SUMMARY:
A tumoral obstruction of the main stem bronchus is frequently observed in the follow-up of lung cancers with a high impact on survival and quality of life of these patients. The endoluminal resection of these tumors through interventional bronchoscopy can remove the tumor but fails to prevent the recurrence. A stent insertion could achieve this goal but this option was never proved in a prospective protocol.

The aim of this study is to analyze the impact of stent insertion on the survival without symptoms of bronchial obstruction in patients treated for their cancer with and without a first line treatment (chemo-radiotherapy or chemotherapy). The patients will be included after resection of the endoluminal symptomatic tumoral obstruction. We will test the effect of the silicone stent insertion ( from NovatechR ) by comparing a stent arm (170 patients with stent insertion) with a control arm (170 patients without stent). The inclusion period will last 3 years with one year of follow-up for each patient. The one-year survival without symptomatic recurrence (proved on bronchoscopy with more than 50% of obstruction in the treated zone) will be the main endpoint. All patients without symptomatic recurrence at one year will be controlled endoscopically. Survival and stent tolerance will be studied as secondary endpoints. All endoscopic events will be depicted on photographs or videos. Each endoscopical situation (before and after resection, recurrence or side effects of stents) will be analyzed and registered by an independent committee of 3 international experts.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years
* non-small cell lung cancer,
* inoperable and location : tracheal, carinal, main bronchus right or left, or intermediate trunk.
* TNM stage known and oncological treatment later determined
* central initial intrinsic bronchial obstruction > 50%.
* resection of tumor with endoscopy, to obtain after therapeutic bronchoscopy a diameter > 50% normal diameter of bronchial segment achieved.
* Tumoral segment fully recoverable by a stent
* Written consent, free and informed
* Patient affiliated or who is entitled to to a social security scheme.

Exclusion Criteria:

* against-indication for general anesthesia.
* Patient with one lung not working beyond the stenosis
* Patient under guardianship
* Pregnancy
* 12 months follow-up impossible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2008-11; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Death and / or symptomatic recurrence (proved on bronchoscopy with more than 50% of obstruction in the treated zone) | 12 months

SECONDARY OUTCOMES:
death | 12 months
For patients who had no symptomatic recurrence of bronchial obstruction Presence of a bronchial stenosis> 50% on a systematic bronchial endoscopy months. | 12 months
Complications of symptomatic trachea-bronchial prosthesis (mobility or migration, granuloma, congestion) motivating endoscopy. | 12 months
Quality of life : EORTC | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Michel Vergnon, MD PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (13):
- France (13):
  - Department of pneumology, CHU Amiens, Amiens
  - Departement of pneumology, CHU Brest, Brest
  - Pneumology departement, Hôpital Percy, Clamart
  - Pneumology departement, CHRU Lille, Lille
  - Pneumology departement, CHU Limoges, Limoges
  - Pneumology departement, Sainte Marguerite hospital, Marseille
  - Pneumology departement, CHU Nantes, Nantes
  - Pneumology departement, Saint-Antoine hospital, Paris
  - Department of respiratory diseases and allergic, Thoracic Oncology, CHU Reims, Reims
  - Pneumology Clinic - Albert Calmette hospital- CHU Rouen, Rouen
  - Pneumology departement CHU Saint-Etienne, Saint-Etienne
  - Endoscopy unit, Thoracic surgery department, Foch Hospital, Suresnes
  - Departement of pneumology, CHU TOULOUSE, Toulouse